CLINICAL TRIAL: NCT06976086
Title: A Prospective, Multicenter, Single-arm Clinical Investigation of the Safety and Performance of the Sentio System in a Pediatric Population
Brief Title: Pediatric Expansion Study of the Sentio System
Acronym: BC119
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); Birmingham Women's and Children's NHS Foundation Trust (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); University Medical Center Groningen (Other); Radboud University Medical Center (Other); Hospital Universitario La Fe (Other); Hospital Universitario Virgen Macarena (Other); Hospital Donostia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC119; CIV-4-12-050315 (Other: EUDAMED); CI/2024/0074/GB (Other: MHRA)
Record Dates: First submitted 2025-04-25; First posted 2025-05-16 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Hearing Loss, Conductive; Hearing Loss, Mixed; Single Sided Deafness
Keywords: Sentio system; Paediatric; Hearing loss; Children; Bone conduction; Transcutaneous
MeSH Terms: conditions — Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural; Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sentio system (Experimental): Prospective, open label, single-arm multicentre investigation designed to follow clinical practice for bone conduction devices.
  Interventions: Device: Active transcutaneous bone conduction system

INTERVENTIONS:
Device: Active transcutaneous bone conduction system — The Sentio system consists of the Sentio 1 Mini sound processor (SP) and Sentio Ti implant with fixation band and screws.
  Other Names: Sentio system

SUMMARY:
This study is performed to collect safety and performance data supporting the use of the Sentio system in children below 12 years of age. The system is currently available on the market for patients 12 years and above. It is a prospective study conducted at eight European hospitals, aiming to treat 50 patients with a hearing loss than would benefit from treatment with a bone-anchored hearing system (BAHS). The primary objective of the study is to demonstrate that the Sentio system improves the hearing on the implanted ear, compared with the unaided situation.

DETAILED DESCRIPTION:
This study is performed to collect safety and performance data supporting the use of the Sentio system in children below 12 years of age. The system is currently available on the market for patients 12 years and above. It is a prospective, multicentre study sponsored by Oticon Medical AB, which will be conducted at eight hospitals across Europe (UK, Spain and the Netherlands). A total of 50 patients with a hearing loss than would benefit from treatment with a bone-anchored hearing system (BAHS) will be included. Participation is voluntary and the decision to participate must be well-founded and well informed.

The Sentio system is a transcutaneous bone conduction hearing system (an implant and an external sound processor) for individuals with certain types of hearing losses. The implant is implanted into the bone behind the ear (mastoid and temporal bone area). After a period of skin healing, a sound processor which transmits sound waves to the implant can be magnetically attached. The implant transforms the sound waves to vibrations, which are then transmitted to the inner ear via the bone. The primary objective of the study is to demonstrate that the Sentio system improves the hearing on the implanted ear, compared with the unaided situation.

The study includes eight study visits; one before surgery, the surgery visit, and six follow-up visits, with the last visit taking place 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form (depending on age of child, signed by parent or legal guardian and child)
2. Subject aged 3 to 11 years
3. Subject with:

   3.1 conductive or mixed hearing losses with pure tone average (PTA) bone conduction (BC) threshold (measured at 0.5, 1, 2 and 3 kHz) of the indicated ear better than or equal to 45 dB HL.

   3.2 OR subject who has a profound sensorineural hearing loss in one ear and normal hearing in the opposite ear (i.e. SSD). The pure tone average (PTA) air conduction (AC) threshold of the hearing ear should then be better than or equal to 20 dB HL (measured at 0.5, 1, 2 and 3 kHz) 3.3 OR subject indicated for an air-conduction contralateral routing of signals (AC CROS) hearing aid, but who for some reason cannot or will not use an AC CROS.
4. Subject and parent or legal guardian have the ability and willingness to comply with investigational procedures/ requirements, as determined by the investigator.
5. Subject with prior experience of amplified sound through a properly fitted hearing aid, a CROS device, or a non-surgical bone anchored solution (e.g. softband).
6. For subject with conductive or mixed hearing losses, ensure sufficient air bone gap (ABG) at the ear to be implanted.
7. Sufficient bone quality/quantity/depth or skull size for implantation of a Sentio Ti implant as assessed according to clinical practice.

Exclusion Criteria:

1. Medical condition that contraindicates implant surgery or anesthesia as judged by the investigator.
2. Untreated ongoing middle ear infection at the time of surgery.
3. Known or suspected contact allergy to silicone or other material used in the Sentio system.
4. Known condition that could jeopardize wound healing and skin condition, e.g. uncontrolled diabetes over time, as judged by the investigator.
5. Known skin or scalp conditions that may preclude attachment or interfere with the usage of the sound processor.
6. Evidence of conditions that would prevent good speech recognition potential as determined by good clinical judgment.
7. Any other known condition that the investigator determines could interfere with compliance or investigation assessments.
8. Use of ototoxic drugs that could be harmful to the hearing, as judged by the investigator.
9. Subject that has received radiotherapy in the area of implantation or is planned for such radiotherapy or similar during the investigation period.
10. For bilateral asymmetric candidates, subject already treated with a bone-anchored hearing solution on the side with the best bone conduction thresholds.
11. Known chronic or non-revisable vestibular or balance disorder.
12. Known abnormally progressive hearing loss.
13. Currently participating, or participated within the last 30 days, in another clinical investigation involving an investigational drug or device that could impact the safety or effectiveness of the Sentio system as determined by the investigator.
14. Use of active implantable or body worn device that for medical reasons cannot be removed or discontinued, such as CSF shunts, implantable cardiac pacemakers, defibrillators, or neurostimulators.
15. Known need for frequent MRI investigations for follow-up of other diseases.
16. Any subject that according to the Declaration of Helsinki is deemed unsuitable for investigation enrolment.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Demonstrate that the Sentio system improves hearing on the implanted ear. | 3 months post-surgery
  Functional gain with the Sentio system, i.e. the difference between pre-operative unaided and post-operative aided sound field thresholds on the implanted ear. The functional gain is calculated as the average of frequencies 500, 1000, 2000 and 4000 Hz (PTA4).

SECONDARY OUTCOMES:
Evaluation of the safety profile of the Sentio system in terms of the occurrence of adverse events and serious adverse events related to the device. | 3 months post-surgery
  Tabulated adverse events and serious adverse events related to the device reported from surgery throughout the investigation reported at 3 months post-surgery.
Functional gain | 12 months post-surgery
  Functional gain is used to assess the performance of the Sentio system. The functional gain is a calculation and is defined as the difference between unaided and aided sound field thresholds. The average functional gain is calculated as the average of frequencies 500, 1000, 2000 and 4000 Hz (PTA4).
Effective gain | 12 months post-surgery
  Effective gain is used to assess the degree the Sentio system compensates for the hearing loss on the implanted ear in patients with mixed/conductive hearing losses. Effective gain is a calculation and is defined as the aided threshold relative to the BC (unmasked bone conduction) threshold and is calculated as the difference in dB between aided sound field thresholds and BC in situ hearing thresholds. The average effective gain (PTA4) is calculated as the average of frequencies 500, 1000, 2000 and 4000 Hz.
Assessment of speech recognition improvement | 3 months post-surgery
  Difference in speech recognition score (%) between pre-operative unaided condition and Sentio-aided condition, measured in quiet on the implanted ear.
Assessment of listening-related fatigue | 6 months post-surgery
  Change in Vanderbilt Fatigue Scale (VFS) questionnaire score between pre-operative unaided condition at baseline and aided condition post-surgery.
  The Vandebilt Fatigue Score questionnaire as a valid measure of listening-related fatigue in children.
Assessment of quality of life | 12 months post-surgery
  Glasgow Children Benefit Inventory (GCBI) questionnaire score addressing the consequences of a specific intervention on various aspects of the child's day-to-day life. The score goes from -100 (max negative effect) to +100 (max positive effect).
Usage hours | 12 months post-surgery
  Sound processor usage hours per day.
Duration of surgery | 3 months post-surgery
  Average length of surgery measured in minutes.
IPS (Inflammation, Pain, Skin numbness) scores | 12 months post-surgery
  Distribution of IPS scores (Inflammation score 0-4; Pain score 0-2; Skin numbness score 0-2) assigned by investigator. The IPS score is presented as [Ix Px Sx] with x being the individual score for each parameter. A higher score corresponds to a poorer outcome.

CONTACTS AND LOCATIONS:
Locations (8):
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Radboud University Medical Center, Nijmegen
- Spain (3):
  - Hospital Universitario de Donostia, San Sebastián
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario y Politécnico La Fe, Valencia
- United Kingdom (3):
  - Birmingham Children's hospital, Birmingham Women's and Children's NHS Foundation Trust, Birmingham
  - The Evelina London Children's Hospital, Guy's and St Thomas' NHS Foundation Trust, London
  - Great Ormond Street Hospital, Great Ormond Street Hospital for Children NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No